CLINICAL TRIAL: NCT03343678
Title: An Open-label, Multi-centre, Phase Ib Trial to Determine the Dose of Intravenous BI 836826 in Combination With Oral Venetoclax in Chronic Lymphocytic Leukaemia Patients Who Are Eligible for Treatment With Venetoclax
Brief Title: This Study in Patients With Chronic Lymphocytic Leukaemia is Done to Determine a Safe and Effective Dose of BI 836826 in Combination With Venetoclax
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Company strategic decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1270.13; 2014-004957-16 (EudraCT Number)
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax; BI 836826

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax + BI 836826 (Experimental)
  Interventions: Drug: Venetoclax; Drug: BI 836826

INTERVENTIONS:
Drug: Venetoclax — Venetoclax given alone and then in combination with BI 836826
Drug: BI 836826 — Venetoclax given in combination with BI 836826

SUMMARY:
The main objective of this trial is to determine the maximum tolerated dose (MTD) of BI 836826 in combination with venetoclax on the basis of dose limiting toxicities (DLTs incidence rate during the MTD evaluation period of the combination treatment and to determine the recommended Phase II dose (RP2D) of the combination.

Other objectives are to evaluate the pharmacokinetics of BI 836826 in combination with venetoclax and to further determine the safety, as well as to evaluate the efficacy of the combination by means of the Complete Response (CR) rate and Minimal Residual Disease (MRD) negativity rate.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Chronic Lymphocytic Leukaemia (CLL) according to International Workshop for Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria documented in medical records
* Indication for treatment of CLL based on investigator's assessment consistent with accepted IWCLL criteria
* Relapsed or refractory CLL after standard therapy in line with the following requirements:

  * Presence of TP53 (Tumour Protein) mutation or deletion (17p), AND at least one prior therapy for CLL with a B-cell receptor pathway inhibitor or contra-indication to the prescription of a B-cell receptor pathway inhibitor OR
  * Absence of TP53 mutation or deletion (17p) AND at least 2 prior treatment regimens for CLL including:

    * at least 4 cycles of chemo-immunotherapy containing a CD20-targeting monoclonal antibody, i.e. at least 4 doses of a monoclonal antibody and at least 4 doses of a cytotoxic AND
    * a B-cell receptor pathway inhibitor
* Clinically quantifiable disease burden defined as

  * either Absolute Lymphocyte Count (ALC) >10x10^9/L, or
  * measurable lymphadenopathy (at least one node > 2 cm on Computed Tomography (CT) scan) or
  * quantifiable bone marrow infiltration documented in a bone marrow biopsy during screening if applicable
* Resolution of all clinically relevant acute non-hematologic toxic effects of any prior antitumour therapy to Grade <=1 with the exception of alopecia or neurotoxicity (Grade 1 or 2 neurotoxicity permitted) prior to the first dose of venetoclax
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2
* Patient of full age (according to local legislation, usually >= 18 years) at screening.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per International Conference on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion criteria:

* Known transformation of Chronic Lymphocytic Leukaemia (CLL) to an aggressive B-cell malignancy at the time of screening (e.g. large B-cell lymphoma, Richter's syndrome)
* History of a non-CLL malignancy except for the following:

  * adequately treated local basal cell or squamous cell carcinoma of the skin,
  * cervical carcinoma in situ,
  * superficial bladder cancer,
  * asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for >=1 year prior to enrolment,
  * other adequately treated Stage 1 or 2 cancer currently in complete response,
  * or any other cancer that has been in complete response for >=2 years.
* Ongoing systemic immunosuppressive therapy other than corticosteroids
* Previous treatment with a CD37-targeting antibody or antibody drug conjugate
* Absolute neutrophil count < 1 x 10^9/L
* Platelet count < 50 x 10^9/L
* Aspartate Transaminase (AST) and/or Alanine Transaminase (ALT) > 3 times the upper limit of normal (ULN) range
* Bilirubin > 1.5 time ULN range with the exception of known Gilbert's syndrome
* Estimated glomerular filtration rate (GFR) <30 mL/min/1.73m2 (based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula)
* Human Immunodeficiency virus (HIV) infection
* Active hepatitis B infection (defined as presence of Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA). (Note: Laboratory tests performed as routine procedure prior to signing ICF but within 2 weeks prior to Cycle 1 Day 1 may be used).
* Cytomegalovirus (CMV) viraemia (Note: Laboratory tests performed as routine procedure prior to signing Informed Consent Form (ICF) but within 2 weeks prior to Cycle 1 Day 1 may be used).
* Active bacterial, viral, or fungal infection requiring systemic treatment.
* Other concomitant clinically significant illness, medical condition, surgical history, physical finding, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia requiring therapy (with the exception of extrasystoles or minor conduction abnormalities), Electrocardiogram (ECG) finding, or laboratory abnormality that in the investigator's opinion could potentially adversely affect the safety of the patient or impair the assessment of trial results
* Known or suspected hypersensitivity to the trial medications or excipients
* Known allergy to xanthine oxidase inhibitors and/or rasburicase in patients at risk of Tumour Lysis Syndrome (TLS)
* Prior treatment with a BCL2i (B-Cell Lymphoma-2 protein) unless the patient has started venetoclax treatment and is still in the ramp-up phase
* Use of a strong CYP3A inhibitor (e.g., ketoconazole, ritonavir, clarithromycin, itraconazole, voriconazole, posaconazole) or of a moderate CYP3A inhibitor (e.g., erythromycin, ciprofloxacin, diltiazem, fluconazole, verapamil), use of a strong CYP3A inducer (e.g., carbamazepine, phenytoin, rifampicin) or a moderate CYP3A inducer (e.g., bosentan, efavirenz, etravirine, modafinil, nafcillin) within five times the half-life of the drug before the initiation of the venetoclax ramp-up period
* Use of a Permeability GlycoProtein (P-gp) inhibitor (e.g., rifampicin) or a breast cancer resistance protein (BCRP) inhibitor within five times the half-life of the drug before the initiation of the venetoclax ramp-up period
* Women who are pregnant, breastfeeding, or who plan to become pregnant while in the trial
* Patients unable to comply with protocol
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Patients who are under judicial protection and patients who are legally institutionalized
* Concomitant participation to a non-CLL investigational device or drug trial or within 30 days after end of participation
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-17 (Estimated); Primary Completion 2018-05-25 (Estimated); Study Completion 2020-11-25 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) based on the number of patients with dose limiting toxicities (DLTs) in the MTD evaluation period | up to 28 days
Number of patients with dose limiting toxicities (DLTs) in the Maximum tolerated dose (MTD) evaluation period | up to 28 days

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve at steady-state (AUCtau) of BI 836826 when administered in combination with venetoclax with an observation time of 28 days in Cycle 1 of the combination. | up to 28 days
Complete response (CR) defined by investigator's assessment based on response assessment at imaging time points, analysed by complete response rate | up to 36 months
Minimal residual disease (MRD) negativity based on blood and analysed by MRD negativity rate | up to 36 months
Minimal residual disease (MRD) negativity based on bone marrow and analysed by MRD negativity rate | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim